CLINICAL TRIAL: NCT00005641
Title: T-Cell Depletion for Graft-Versus-Host Disease (GVHD) Prevention in High Risk Matched and Mismatched Allogeneic Bone Marrow Transplantation
Brief Title: Removal of T Cells to Prevent Graft-Versus-Host Disease in Patients Undergoing Bone Marrow Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low study accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 11587; MCC-11587; MCC-IRB-4599; NCI-G00-1781; BB-IDE-7181 (Other: FDA)
Record Dates: First submitted 2000-05-02; First posted 2004-06-08 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; refractory multiple myeloma; stage 0 chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Leucovorin; Methotrexate; Methylprednisolone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: leucovorin calcium
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Eliminating the T cells from the donor cells before transplanting them may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of T cell removal to prevent graft-versus-host disease in patients who are undergoing bone marrow transplantation from a donor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the incidence and severity of graft vs host disease (GVHD) following allogeneic bone marrow transplantation with marrow grafts modified by T cell depletion with counterflow centrifugal elutriation and CD34+ cell selection in patients at high risk for GVHD. II. Determine the incidence of graft failure following this treatment regimen in this patient population. III. Determine the relapse rate and overall survival in this patient population treated with this regimen.

OUTLINE: Patients with unrelated donors, mismatched related donors, or matched related donors diagnosed with acute lymphocytic leukemia, chronic lymphocytic leukemia, myeloma, or advanced acute myeloid leukemia (AML), receive cyclophosphamide IV over 60 minutes on days -6 and -5 and fractionated total body irradiation (TBI) 3 times a day on days -3 through -1, and twice on day 0. Patients receive graft vs host disease (GVHD) prophylaxis with anti-thymocyte globulin (ATG) IV over 8 hours on days -2 and -1. Patients undergo allogeneic bone marrow transplantation (ABMT) on day 0 with marrow grafts modified by T cell depletion with counterflow centrifugal elutriation and CD34+ selection. Patients unable to receive TBI due to matched or mismatched related donors, or age (56 to 60), or patients diagnosed with AML-CR1, chronic myelogenous leukemia, myelodysplastic syndrome, or myeloproliferative disorders with matched related donors, receive oral busulfan every 6 hours on days -7 through -4, cyclophosphamide IV over 60 minutes on days -3 and -2, and ATG IV over 8 hours on days -2 and -1 for GVHD prophylaxis. Patients undergo T cell depleted ABMT on day 0. At pretransplantation, patients with acute leukemia receive intrathecal (IT) methotrexate (MTX) following lumbar puncture. At 48 hours following IT MTX, patients with CNS involvement receive a second dose of IT MTX followed by oral leucovorin calcium every 6 hours for 4 doses. Patients with prior CNS involvement receive cranial radiotherapy for 2 weeks. Following AMBT, patients undergo GVHD prophylaxis consisting of methylprednisolone IV every 12 hours on days 5-22, and then once daily on days 23-28 and cyclosporine IV or orally twice daily beginning on day -1 and continuing until 7-9 months following ABMT. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy Acute myeloid leukemia (AML) Complete remission 1 (CR1): high risk defined by poor cytogenetics (e.g., deletions, additions, or multiple abnormalities) Complete remission 2 (CR2) Induction failures Relapse: at least one reinduction attempt if at least 10% marrow blasts Acute lymphocytic leukemia CR1: high risk defined by overt CNS involvement or poor cytogenetics (e.g., additions, deletions, translocations, or multiple abnormalities) CR2 Induction failures Relapse as for AML Chronic myelogenous leukemia Chronic phase (CP) 1 Accelerated phase (AP)/CP2: blast phase patients require induction and achievement of a second chronic phase prior to transplantation Chronic lymphocytic leukemia Relapse: any stage and must have received no greater than 3 regimens since diagnosis Multiple myeloma Primary refractory disease at diagnosis Relapse (no greater than 2): sensitive disease Plasma cell leukemia Inability to achieve a complete remission or relapse after autologous transplantation (no greater than 40 years) Myelodysplasia All FAB subtypes Myeloproliferative disorders Poor response to medical therapy OR Cytogenetic abnormalities Severe aplastic anemia (SAA) (for unrelated and/or mismatched donors) Very SAA at diagnosis OR SAA: induction failures One antigen mismatch (recipient age 15 to 55) Related donors may be A, B, or DR mismatched Unrelated donors may be A or B mismatched (DRB1 match) Phenotypic (6 out of 6) match Recipient age 51 to 60 if related donor Recipient age 41 to 55 if unrelated donor

PATIENT CHARACTERISTICS: Age: 15 to 60 Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT/SGPT no greater than 3 times normal PT/PTT normal Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: LVEF at least 45% by MUGA scan or echocardiography Greater than 6 months since myocardial infarction No uncontrolled arrhythmias Pulmonary: FEV1 and DCLO at least 50% predicted Other: No psychosocial conditions that would preclude study No uncontrolled diabetes mellitus No uncontrolled thyroid disease No active serious infections HIV negative Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1997-09; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Goldstein, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States